CLINICAL TRIAL: NCT04797780
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of Tamibarotene Plus Azacitidine Versus Placebo Plus Azacitidine in Newly Diagnosed, Adult Patients Selected for RARA-positive Higher-risk Myelodysplastic Syndrome (SELECT MDS-1)
Brief Title: Tamibarotene Plus Azacitidine in Participants With Newly Diagnosed RARA-positive Higher-Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As per Sponsor decision, the study was terminated.
Sponsor: Syros Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY-1425-301; 2020-004528-40 (EudraCT Number)
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Higher-Risk; Retinoic Acid Receptor Alpha (RARA) positive; Newly Diagnosed; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — tamibarotene; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tamibarotene + Azacitidine (Experimental): Tamibarotene: 6 mg administered orally twice per day (BID) on Days 8 through 28 of each 28-day treatment cycle.
  Azacitidine: 75 mg/m^2 administered intravenously or subcutaneously each day on Days 1 through 7 of each 28-day treatment cycle.
  Interventions: Drug: Tamibarotene; Drug: Azacitidine
- Tamibarotene Matched Placebo + Azacitidine (Placebo Comparator): Placebo: Tamibarotene-matching tablets administered orally BID on Days 8 through 28 of each 28-day treatment cycle.
  Azacitidine: 75 mg/m^2 administered intravenously or subcutaneously each day on Days 1 through 7 of each 28-day treatment cycle.
  Interventions: Drug: Placebo; Drug: Azacitidine

INTERVENTIONS:
Drug: Tamibarotene — Administered as specified in the treatment arm
  Other Names: SY-1425
  Arms: Tamibarotene + Azacitidine
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Tamibarotene Matched Placebo + Azacitidine
Drug: Azacitidine — Administered as specified in the treatment arm

SUMMARY:
This study compares the efficacy of Tamibarotene in combination with azacitidine to azacitidine in combination with placebo in participants who are Retinoic Acid Receptor Alpha (RARA) positive, and newly diagnosed with higher-risk myelodysplastic syndrome (HR-MDS), and who have not received treatment for this diagnosis. The primary goal of the study is to compare the complete remission rate between the two treatment arms.

DETAILED DESCRIPTION:
A subset of participants have MDS characterized by an overexpression of the RARA gene. A blood test will be used to identify participants with RARA-positive MDS. Assessment of the RARA biomarker for study eligibility will be done by collection of blood samples from potential study participants at the pre-screening visit and testing at a central laboratory. Participants who meet eligibility requirements will be randomized 2:1 to receive either Tamibarotene plus azacitidine or placebo plus azacitidine.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be RARA-positive based on the investigational assay.
* Participants must be newly diagnosed with HR-MDS as follows:

  * Diagnosis of MDS according to the World Health Organization (WHO) classification and classified by the Revised International Prognostic Scoring System (IPSS R) risk category as very high, high, or intermediate risk.
* Participants must have Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.

Key Exclusion Criteria:

* Participants are suitable for and agree to undergo allogeneic hematopoietic stem cell transplant (HSCT) at the time of screening.

  * Participants who need treatment prior to stem cell transplant can receive treatment on this study and stop the study treatment when they are ready to proceed to transplant.
* Participants who received prior treatment for MDS with any hypomethylating agent, lenalidomide, chemotherapy or allogeneic HSCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Syros Pharmaceuticals Inc.
Locations (128):
- United States (22):
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - University of California, Los Angelas, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Comprehensive Hematology and Oncology, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tulane Cancer Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Morristown Medical Center- Atlantic Hematology Oncology, Morristown, New Jersey
  - Northwell Health, Lake Success, New York
  - Novant Health Inc, Charlotte, North Carolina
  - Novant Health Cancer Institute - Forsyth, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - TriStar - Sarah Cannon BMT, Nashville, Tennessee
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington
- Austria (3):
  - Medical University of Graz, Graz
  - Salzburg Cancer Research Institute (SCRI), Salzburg
  - Klinik Hietzing, Vienna
- Belgium (7):
  - ZNA Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Ghent University Hospital, Ghent
  - Hospital De Jolimont, La Louvière
  - CHU de Liège, Liège
  - AZ Delta, Roeselare
  - CHU-UCL Namur, Yvoir
- Canada (7):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Tom Baker Cancer Centre, Calgary
  - London Health Sciences Centre, London
- Czechia (3):
  - Fakultni nemocnice Olomouc (University Hospital Olomouc), Olomouc
  - University Hospital Ostrava, Ostrava
  - General University Hospital Prague, Prague
- France (20):
  - CHU Amiens-Picardie, Amiens
  - CHU d'Angers, Angers
  - Centre Hospitalier de la Côte Basque Hématologie Clinique, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHRU de BREST - Hôpital Morvan, Brest
  - CHU Clermont Ferrand / CHU Estaing, Clermont-Ferrand
  - CHU Grenoble Alpes Hôpital Nord Michallon, La Tronche
  - Hopital Mignot, Le Chesnay
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CHU la Conception, Marseille
  - CHU Nantes - Hotel Dieu, Nantes
  - CHU de Nice - Hopital L'Archet, Nice
  - Hôpital Saint Louis, Paris
  - CHU Bordeaux, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Poiters, Poitiers
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - ICANS Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Universitätsklinikum Augsburg, Augsburg
  - Helios Klinikum Berlin Buch GmbH, Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Marburg, Marburg
  - Universitätsklinikum Münster, Münster
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Debrecen University Medical and Health Science Centre, Debrecen
  - Markhot Ferenc Oktatókórház és Rendelőintézet, Belgyógyászati- és Infektológiai Centrum, Eger
  - Petz Aladar County Teaching Hospital, Győr
  - Josa Andras Teaching Hospital, Nyíregyháza
- Israel (6):
  - Barzilai Medical Center of Ashkelon, Ashkelon
  - Bnai Zion Medical center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - AOU Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - Romagnolo Institute to Study Tumors "Dino Amadori "/ Meldona, Meldola
  - A.O.U. Maggiore della Carità, Novara
  - Ospedali Marche Nord Centro Ematologia e Trapianti, Pesaro
  - Ospedale S.Maria delle Croci, Ravenna
  - Ospedale S. Eugenio - ASL Roma 2, Roma
  - Fondazione Policlinico Tor Vergata, Rome
  - AOUI di Verona, Verona
- Poland (6):
  - University Clinic Gdansk, Gdansk
  - Pomeranian Hospital Gdynia, Gdynia
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
  - University Clinic Warsaw, Warsaw
  - Alfred Sokołowski Hospital Wałbrzych, Wałbrzych
- Spain (22):
  - Institut Catala d'Oncologia - Hospital Duran i Reynals Location, Badalona
  - Hospital del Mar, Barcelona
  - H. Santa Creu i Sant Pau, Barcelona
  - Fundación Privada Instituto de Investigación Oncológica Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar Secretaria d'Hematologia Clínica, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - H. Universitario La Paz, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturia, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Clinica Universidad Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (8):
  - Castle Hill Hospital, Cottingham, Cottingham
  - Ninewells Hospital, Dundee
  - Western General Hospital in NHS Lothian Edinburgh Scotland, Edinburgh
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - King's College Hospital NHS Foundation Trust, London
  - The Royal Marsden Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Sandwell and West Birmingham Hospital NHS Trust, West Bromwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeZern AE, Thepot S, de Botton S, Patriarca A, Deeren D, Torregrossa-Diaz JM, Marconi G, Bernal T, Bergua Burgues J, Xicoy B, Jonasova A, Zeidan AM, Dimicoli-Salazar S, Simand C, Valcarcel D, Diez Campelo M, Chai-Ho W, Saini L, Garnier A, Geissler K, Ofran Y, Nagy Z, Krishnamurthy P, Lubbert M, Basak G, Carraway HE, Sallman DA, Borate U, Santini V, Campbell V, Fenaux P, Braun T, Lanza F, Zaucha JM, Roth DA, Paul S, Roy P, Kelly MJ, Volkert A, Chisholm J, Malak TA, Klimek VM, Cluzeau T. Pivotal results of SELECT-MDS-1 phase 3 study of tamibarotene with azacitidine in newly diagnosed higher-risk MDS. Blood Adv. 2025 Aug 26;9(16):4090-4099. doi: 10.1182/bloodadvances.2025016229. PMID 40334070
- [Derived] Stahl M, DeZern AE. Is there a path forward for immunotherapy in patients with myelodysplastic syndromes? Lancet Haematol. 2024 Jan;11(1):e5-e7. doi: 10.1016/S2352-3026(23)00343-5. Epub 2023 Dec 5. No abstract available. PMID 38065202

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per Sponsor decision, the study was terminated. Number of participants who started and completed the study and reasons for study discontinuation were collected for the Intent-To-Treat (ITT) analysis set and included all participants who were randomized; data were collected by study arm regardless of the dose level received.
Groups:
- Tamibarotene + Azacitidine: Tamibarotene: 6 milligrams (mg) administered orally twice per day (BID) on Days 8 through 28 of each 28-day treatment cycle. Azacitidine: 75 mg/meter square (m^2) administered intravenously or subcutaneously each day on Days 1 through 7 of each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Started (ITT Analysis set.) | 164 | 82
Modified Intent to Treat (mITT) Analysis Set (The mITT analysis set included the first approximately 190 randomized participants.) | 126 | 64
Safety Analysis Set 1 (The Safety Analysis Set 1 included all participants who were randomized and had received any amount of study drug (tamibarotene, placebo, or azacitidine); data were collected by dose level received.) | 160 | 85
Completed | 100 | 52
Not Completed | 64 | 30
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 14 | 9
Not completed — Death | 49 | 20

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were collected for the ITT Analysis Set and included all participants who were randomized; data were collected by study arm regardless of the dose level received.
Groups:
- Tamibarotene + Azacitidine: Tamibarotene: 6 mg administered orally BID on Days 8 through 28 of each 28-day treatment cycle. Azacitidine: 75 mg/m^2 administered intravenously or subcutaneously each day on Days 1 through 7 of each 28-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine | Total
Number analyzed (Participants) | 164 | 82 | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 7 | 22
  >=65 years | 149 | 75 | 224
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 21 | 71
  Male | 114 | 61 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 58 | 35 | 93
  Unknown or Not Reported | 102 | 47 | 149
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 58 | 31 | 89
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 101 | 49 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission (CR)
Description: CR was determined by the investigator per the modified International Working Group Myelodysplastic Syndrome (IWG MDS). CR was defined as participants with hemoglobin ≥11 grams/deciliter (g/dL), neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, bone marrow blasts (BMBs) ≤5% and normal maturation of all cell lines, persistent dysplasia were noted.
Time Frame: Up to 45 months
Population: The mITT analysis set included the first approximately 190 randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 126 | 64
Percentage of participants | 23.81 [16.7 to 32.2] | 18.75 [10.1 to 30.5]
Statistical Analysis 1: Comparison: Tamibarotene + Azacitidine vs Tamibarotene Matched Placebo + Azacitidine; Test type: Superiority; p = 0.2084, Cochran-Mantel-Haenszel; Difference in CR Rate = 5.060, 95% CI 2-sided [-7.1 to 17.2]

2. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR: duration from date of first documented evidence of CR, partial remission (PR), marrow CR (mCR), or hematologic improvement (HI) to date of documented disease progression or relapse of disease as determined by investigator per modified IWG MDS criteria or death due to any cause, whichever occurred first. CR: hemoglobin (Hb)≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs≤5% & normal maturation of all cell lines, persistent dysplasia. PR: Hb ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs decreased by ≥50% from baseline, but >5%. mCR: Hb ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs decreased by≥50% from baseline, & ≤5%. Subcategories of HI included erythroid response (Hgb increase by ≥1.5 g/dL), platelet response (absolute increase of≥30*10^9/L if starting with >20*10^9/L platelets; increase from <20 to >20*10^9/L and by ≥100%),neutrophil response (≥100% increase & absolute increase >0.5*10^9/L).
Time Frame: Up to 45 months
Population: The mITT analysis set included the first approximately 190 randomized participants. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 35 | 16
Months | 12.0 [7.9 to 22.1] | 19.4 [5.8 to NA] — The upper limit of 95% confidence interval (CI) could not be calculated due to not enough participants with an event.

3. Secondary Outcome: Number of Participants Who Achieved Transfusion Independence (TI)
Description: TI was defined as a period of at least 56 days with no red blood cell (RBC) or platelet transfusion since the date of randomization to the last dose of study drug + 30 days, the initiation of post-treatment therapy, or death, whichever occurred first.
Time Frame: Up to 45 months
Population: The mITT analysis set included the first approximately 190 randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 126 | 64
Participants | 85 | 38

4. Secondary Outcome: Percentage of Participants Who Achieved Overall Response (OR)
Description: OR: Participants who achieved CR, PR, mCR, or subcategories of HI, as determined by investigator per modified IWG MDS criteria. CR was defined as hemoglobin ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, bone marrow blasts (BMBs) ≤5% and normal maturation of all cell lines, persistent dysplasia were noted. PR was defined as hemoglobin ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs decreased by ≥50% from baseline, but >5%. mCR was defined as hemoglobin ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs decreased by ≥50% from baseline, and ≤5%. Subcategories of HI included erythroid response (Hgb increase by ≥1.5 g/dL), platelet response (absolute increase of ≥30*10^9 /L if starting with >20*10^9/L platelets increase from <20*10^9/L to >20*10^9/L and by at least 100%), neutrophil response (at least a 100% increase and an absolute increase >0.5*10^9 /L).
Time Frame: Up to 45 months
Population: The mITT analysis set included the first approximately 190 randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 126 | 64
Percentage of participants | 71.43 [62.7 to 79.1] | 70.31 [57.6 to 81.1]

5. Secondary Outcome: Duration of Complete Response (DOCR)
Description: DOCR was defined as the duration from the date of first documented evidence of CR to the date of documented relapse of disease or disease progression, as determined by the investigator per the modified IWG MDS criteria, or death due to any cause, whichever occurred first. CR was defined as participants with hemoglobin ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs ≤5% and normal maturation of all cell lines, persistent dysplasia were noted. Among CR responders, DOCR was calculated as: DOCR (months) = (first date of documented relapse of disease, disease progression, or death due to any cause - date of first documented evidence of CR + 1) / 30.4375.
Time Frame: Up to 45 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 7 | 1
Months | 15.7 [6.9 to NA] — The upper limit of 95% CI could not be calculated due to not enough participants with an event. | NA [16.6 to NA] — Median and the upper limit of 95% CI could not be calculated due to not enough participants with an event.

6. Secondary Outcome: Time to Complete Remission (TCR)
Description: TCR was defined as the duration from the date of randomization to the date of the first documented evidence of CR as determined by the investigator per the modified IWG MDS criteria. Among CR responders, this outcome measure was calculated as: Time to CR= (date of the first documented evidence of CR - date of randomization + 1) / 30.4375. CR was defined as hemoglobin ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, bone marrow blasts ≤5% and normal maturation of all cell lines, persistent dysplasia were noted.
Time Frame: Up to 45 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 30 | 12
Months | 4.845 [0.95 to 7.92] | 3.595 [1.38 to 5.88]

7. Secondary Outcome: Time to Initial Response (TIR)
Description: TIR: duration from date of randomization to the date of first documented evidence of CR, PR, mCR, or HI as determined by investigator per modified IWG MDS criteria. CR: hemoglobin (Hb) ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, bone marrow blasts (BMBs) ≤5% and normal maturation of all cell lines, persistent dysplasia. PR: Hb ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs decreased by ≥50% from baseline, but >5%. mCR: Hb ≥11 g/dL, neutrophils ≥1.0*10^9/L, platelets ≥100*10^9/L, blasts 0%, BMBs decreased by ≥50% from baseline, and ≤5%. Subcategories of HI included erythroid response (Hgb increase by ≥1.5 g/dL), platelet response (absolute increase of ≥30*10^9/L if starting with >20*10^9/L platelets increase from <20 to >20*10^9/L and by at least 100%), neutrophil response (at least a 100% increase and absolute increase>0.5*10^9 /L).
Time Frame: Up to 45 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 90 | 45
Months | 1.050 [0.33 to 9.20] | 1.120 [0.72 to 8.61]

8. Secondary Outcome: Change in Health-Related Quality of Life (HRQoL) as Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 Scale (EORTC QLQ-30)
Description: HRQoL was evaluated by EORTC QLQ-C30 global health status/quality of life composite scale in all randomized participants. The QLQ-30 is a cancer-specific, self-administered questionnaire that contains 30 questions, covering global, functional, and symptom scales. Scores range from 0 to 100. Higher scores on global and functional scales indicated better quality of life (QoL), while higher scores on the symptom scales indicated declining QoL.
Time Frame: Up to 45 months
Population: While the QLQ-30 questionnaire was completed to derive data for the planned EORTC QLQ-30 outcome measure, the study was terminated prior to that data from the questionnaire were collected, analyzed, summarized, or made available by the study sponsor. Therefore, no questionnaire data can be presented here.
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in HRQOL as Assessed by the European Quality of Life 5 Dimensions Scale (EuroQoL-5D)
Description: The EQ-5D-3L essentially consisted of- the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprised of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 3 levels: no problems, some problems, extreme problems. Total scale range for each dimension reported was 1 to 3. The EQ VAS recorded the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents. Total scale range for VAS dimension reported was 0 to 100.
Time Frame: Up to 45 months
Population: While the Q-5D-3L questionnaire was completed to derive data for the planned EuroQoL-5D outcome measure, the study was terminated prior to that data from the questionnaire were collected, analyzed, summarized, or made available by the study sponsor. Therefore, no questionnaire data can be presented here.
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence that developed or worsened in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. TEAEs are defined as those AEs with onset after the first dose of study drug or existing events that worsened after the first dose during the study up until the last dose of study drug + 30 days. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 45 months
Population: Adverse Event data were collected for the Safety Analysis Set 1 and included all participants who were randomized and had received any amount of study drug (tamibarotene, placebo, or azacitidine); Adverse Event data were collected by dose level received.
Measure: Count of Participants; unit: Participants
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
Number analyzed (Participants) | 160 | 85
Participants
  TEAEs | 153 | 81
  SAEs | 87 | 32

ADVERSE EVENTS:
Time Frame: Up to 45 months
Description: Data for All-Cause Mortality were collected for the ITT Analysis Set and included all participants who were randomized; data were collected by study arm regardless of the dose level received. Adverse Event data were collected for the Safety analysis set 1 and included all participants in the ITT analysis set who had received any amount of study drug (tamibarotene, placebo, or azacitidine); data were collected by dose level received.
Arm/Group | Tamibarotene + Azacitidine | Tamibarotene Matched Placebo + Azacitidine
All-Cause Mortality (participants affected / at risk) | 49/164 | 20/82
Serious Adverse Events (participants affected / at risk) | 87/160 | 32/85
Other Adverse Events (participants affected / at risk) | 152/160 | 80/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamibarotene + Azacitidine (N=160) | Tamibarotene Matched Placebo + Azacitidine (N=85)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 23 | 10
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 4
Abscess limb (Infections and infestations) | 1 | 0
Achromobacter infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 3 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Legionella infection (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 17 | 5
Pneumonia aspiration (Infections and infestations) | 2 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 3
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pseudomonas test positive (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cranial nerve disorder (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0
Vascular disorders Arteriosclerosis (Vascular disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 2
Bursitis infective (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tamibarotene + Azacitidine (N=160) | Tamibarotene Matched Placebo + Azacitidine (N=85)
Anaemia (Blood and lymphatic system disorders) | 49 | 29
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 3
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 48 | 26
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 18
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 4
Atrial flutter (Cardiac disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Chalazion (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 1
Conjunctival suffusion (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 4 | 0
Eye haematoma (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Scleral haemorrhage (Eye disorders) | 0 | 1
Trichiasis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 3 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 2
Anal inflammation (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 65 | 36
Dental caries (Gastrointestinal disorders) | 0 | 1
Dental discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 32 | 16
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3
Gingival bleeding (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 7 | 2
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia teeth (Gastrointestinal disorders) | 1 | 0
Ileal ulcer (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 43 | 18
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral blood blister (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 9 | 3
Toothache (Gastrointestinal disorders) | 2 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 21 | 12
Administration site erythema (General disorders) | 0 | 1
Asthenia (General disorders) | 50 | 13
Catheter site erythema (General disorders) | 1 | 0
Catheter site irritation (General disorders) | 1 | 0
Catheter site pruritus (General disorders) | 1 | 0
Catheter site rash (General disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 4 | 2
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 16 | 8
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 1
Generalised oedema (General disorders) | 2 | 0
Hyperpyrexia (General disorders) | 1 | 0
Implant site erythema (General disorders) | 1 | 0
Inflammation (General disorders) | 4 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site bruising (General disorders) | 2 | 1
Injection site erythema (General disorders) | 6 | 8
Injection site haematoma (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Injection site pain (General disorders) | 4 | 6
Injection site pruritus (General disorders) | 0 | 3
Injection site rash (General disorders) | 2 | 0
Injection site reaction (General disorders) | 10 | 3
Injection site urticaria (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 4 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 15 | 8
Pain (General disorders) | 3 | 1
Peripheral swelling (General disorders) | 2 | 1
Puncture site pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 41 | 9
Systemic inflammatory response syndrome (General disorders) | 1 | 1
Temperature regulation disorder (General disorders) | 2 | 0
Thirst (General disorders) | 0 | 1
Xerosis (General disorders) | 1 | 0
Biliary cyst (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 3 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 14 | 3
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 2
Chronic sinusitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 0 | 1
Cystitis bacterial (Infections and infestations) | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 4 | 0
Folliculitis (Infections and infestations) | 5 | 2
Folliculitis genital (Infections and infestations) | 0 | 1
Fungal foot infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Genital herpes (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 2 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Hordeolum (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Infective glossitis (Infections and infestations) | 1 | 0
Infestation (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 1
Klebsiella urinary tract infection (Infections and infestations) | 3 | 0
Laryngitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 5 | 1
Oral fungal infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 2 | 2
Oropharyngeal candidiasis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Perineal cellulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 0
Pilonidal disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 3
Pseudomonas infection (Infections and infestations) | 1 | 1
Pulmonary nocardiosis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pustule (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 2 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Rhinovirus infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Systemic mycosis (Infections and infestations) | 1 | 0
Tinea versicolour (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 12 | 3
Varicella (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 4
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 0
Dust inhalation pneumopathy (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 4
Foreign body in ear (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 4 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 8 | 3
Amylase increased (Investigations) | 7 | 1
Aspartate aminotransferase increased (Investigations) | 8 | 1
Blast cell count increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 6 | 3
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 4
Blood calcium decreased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 6 | 1
Blood creatine increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 12 | 3
Blood fibrinogen decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 0
Blood magnesium decreased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 3 | 0
Blood urea increased (Investigations) | 3 | 0
Blood uric acid increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 5 | 1
Cardiac murmur (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 1 | 0
Coagulation time prolonged (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 4 | 3
Enterococcus test positive (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 7 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Heart rate increased (Investigations) | 0 | 1
Human rhinovirus test positive (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 4 | 0
Lipase increased (Investigations) | 4 | 4
Lymphocyte count decreased (Investigations) | 4 | 2
Neutrophil count decreased (Investigations) | 20 | 10
Platelet count decreased (Investigations) | 18 | 13
Prothrombin time prolonged (Investigations) | 1 | 0
Weight decreased (Investigations) | 36 | 5
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 24 | 5
Decreased appetite (Metabolism and nutrition disorders) | 29 | 14
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 4
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 55 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1
Iron overload (Metabolism and nutrition disorders) | 2 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 5
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 12 | 4
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 8 | 2
Dysgraphia (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 11 | 6
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 3
Parkinson's disease (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 3 | 2
Structural brain disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 1
Taste disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 0
Abulia (Psychiatric disorders) | 0 | 1
Acrophobia (Psychiatric disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 8 | 4
Delusion of parasitosis (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Hallucination, visual (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 11 | 1
Mood altered (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 4 | 1
Leukocyturia (Renal and urinary disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urethral prolapse (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/86 | 1/46 — This Adverse event is gender specific. So, the number of participants at risk is male participants only.
Breast pain (Reproductive system and breast disorders) | 1/40 | 0/18 — This Adverse event is gender specific. So, the number of participants at risk is female participants only.
Pelvic pain (Reproductive system and breast disorders) | 2/40 | 0/18 — This Adverse event is gender specific. So, the number of participants at risk is female participants only.
Penile haemorrhage (Reproductive system and breast disorders) | 1/86 | 0/46 — This Adverse event is gender specific. So, the number of participants at risk is male participants only.
Prostatism (Reproductive system and breast disorders) | 0/86 | 1/46 — This Adverse event is gender specific. So, the number of participants at risk is male participants only.
Prostatitis (Reproductive system and breast disorders) | 4/86 | 0/46 — This Adverse event is gender specific. So, the number of participants at risk is male participants only.
Vulvovaginal dryness (Reproductive system and breast disorders) | 2/40 | 0/18 — This Adverse event is gender specific. So, the number of participants at risk is female participants only.
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 8
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Bullous haemorrhagic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0
Mucocutaneous toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pernio-like erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 7
Purpura (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 34 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 2
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 0
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 3 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 12 | 0
Fibromuscular dysplasia (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 6 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 1
Hyperaemia (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 8 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 3
Pallor (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 2 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 4 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 5 | 0
Varicose vein (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
As per Sponsor decision, the study was terminated. Note that the study was terminated prior to the data from the questionnaires were collected, analyzed, summarized, or made available by the study sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Note that the agreements are between the clinical sites and the Sponsor (or its agents), which restrict the clinical trial sites' rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT04797780/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT04797780/SAP_001.pdf